CLINICAL TRIAL: NCT02537067
Title: A Phase III Clinical Trial to Evaluate the Efficacy and Safety of Chondron (Autologus Chondrocyte) in Patients With Cartilage Defects in Their Ankle for 18 Months
Brief Title: Efficacy and Safety of Chondron (Autologus Chondrocyte) in Patients With Cartilage Defects in Their Ankle
Status: Unknown | Phase: Phase 3 | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Sewon Cellontech Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 04CON
Record Dates: First submitted 2015-08-13; First posted 2015-09-01 (Estimated); Last update posted 2015-09-01 (Estimated); Status verified 2015-08

CONDITIONS: Defect of Articular Cartilage; Degenerative Joint Disease of Ankle and/or Foot; Ankle (Ligaments); Instability, Familial
Keywords: a partial cartilage defect of ankle; Chondron; Autologus Chondrocyte

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Autologous cultured Chondrocyte (Experimental): Subjects who give consent will be screened and those who meet trial criteria will receive CHONDRON (Autologous cultured Chondrocyte) by transplant.
  Interventions: Drug: CHONDRON

INTERVENTIONS:
Drug: CHONDRON — 1. Harvesting of ankle or knee cartilage
  2. The cells that fill the vial are sufficiently suspended, and a sufficient amount of suspension is grafted in the defect with fibrin glue.
  Other Names: Autologous cultured Chondrocyte

SUMMARY:
The objective of this study is to evaluate the efficacy and safety of Chondron (Autologus Chondrocyte) in patients with cartilage defects in their ankle for 18 months

DETAILED DESCRIPTION:
This is an open label trial, involving a total of 28 subjects. Subjects who give consent will be screened and those who meet trial criteria will receive CHONDRON (Autologous cultured Chondrocyte) by transplant. During the trial period, subjects must follow the instructions given by principal investigator. Subjects will make 6* hospital visits on a regular basis inclusive of hospitalization. During these visits subjects will be examined. For the evaluation of safety and efficacy of CHONDRON, examination with doctors, x-ray, MRI tests and arthroscopy will be performed. *If tissue samples can be collected at screening visit, there will be only 5 visits.

ELIGIBILITY:
Inclusion Criteria:

* 1. Adult men and women over 15 and less than 65 years of age 2. Applicable to patients who have a partial cartilage defect in their ankle based on an MRI (defect size: for a single lesion, less than 15 cm2; and for multiple lesions, less than 20 cm2) 3. Patients with ankle-tibia malalignment of the ankle joint, unstable ankle ligaments, bone defects at the cartilage defect area or patients who received correction in advance 4. Patients which surrounding cartilage are normal 5.Patients with a Grade III or IV cartilage defect size on the ICRS (International Cartilage Repair Society) 6. Patients who agreed to clinical trial participation voluntarily or by the will of the person in parental authority, and signed the written consent form

Exclusion Criteria:

* 1. Patients hypersensitive to bovine protein 2. Patients hypersensitive to gentamicin antibiotics 3. Patients with inflammatory arthritis such as rheumatoid arthritis, gout arthritis 4. Patients with arthritis related to autoimmune disease 5. Pregnant, breast-feeding patients or those who have a possibility of pregnancy 6. Patients with accompanying diseases other than articular cartilage defects, including tumors 7. Patients who have a history of receiving radiotherapy, chemotherapy in the last 2 years 8. Patients with diabetes (however, patients whose blood sugar test results are normal and do not have any complication of diabetes, when a written opinion that CHONDRON administration is possible is appended by a doctor are excluded) 9. Patients who are administering antibiotics and antimicrobial agents due to infection 10. Patients who receive steroid hormone therapy 11. Patients with psychiatric disorder and those who are considered to be inappropriate for this trial by the judgment of the clinical trial manager

Ages: 15 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 28 (Actual)
Dates: Start 2010-01; Primary Completion 2015-05 (Actual); Study Completion 2015-12 (Estimated)

PRIMARY OUTCOMES:
Grade change of ICRS(International Cartilage Repair Society) by arthroscopy | 12 months after the surgery
  The change of ICRS grade of the affected ankle shall be assessed at 12 months after the surgery. The results on the surgery date shall be considered the baseline data and shall be compared with those at 12 months after the surgery based on arthroscopy. For the final efficacy evaluation, the percentage of the patients (success rate) who showed Grade III or IV ICRS before the surgery and improved to Grade 0 or I after the surgery will be calculated.

SECONDARY OUTCOMES:
Score change of AOFAS(American orthopedic foot & ankle society) Score | baseline and six, 12 and 18 months after the surgery
  The improvements in the AOFAS in the affected ankle at baseline and six, 12 and 18 months after the surgery will be compared. The final efficacy evaluation shall be done by calculating the difference between the AOFAS at the baseline and that 18 months after the surgery.
Hannover Score | baseline and six, 12 and 18 months after the surgery
  The improvements in the Hannover score in the affected ankle at baseline and six, 12 and 18 months after the surgery will be compared. The final efficacy evaluation shall be done by calculating the difference between the Hannover score at the baseline and that 18 months after the surgery.
Score change of Evaluation by physician in charge | six, 12 and 18 months after the surgery
  The improvement will be evaluated by the physician using a five-level scale six, 12 and 18 months after the Chondron grafting.
Score change of 100mmVAS(visual analogue scale) | baseline and six, 12 and 18 months after the surgery
  The improvements of pain in the 100mmVAS in the affected ankle at baseline and six, 12 and 18 months after the surgery will be compared. The final efficacy evaluation shall be done by calculating the difference between the 100mmVAS at the baseline and that 18 months after the surgery.
Comparing MRI results | baseline and 18 months after the surgery
  The morphological improvement from MRI image of the affected ankle will be assessed at 18 months after the surgery from those at baseline. For MRI image at baseline, the MRI should be performed within two weeks from the Chondron grafting for the efficacy evaluation.

CONTACTS AND LOCATIONS:
Overall Officials: Jin Su Kim, MD, Principal Investigator — Eulji General Hospital; Ki Hyuck Sung, MD, Principal Investigator — Myongji Hospital
Locations (2):
- South Korea (2):
  - Myongji Hospital, Goyang-si, Gyeonggi-do
  - Eulji General Hospital, Seoul, Seoul